CLINICAL TRIAL: NCT00882583
Title: A Phase I Study of Dasatinib, Cetuximab and Radiation With or Without Cisplatin in Locally Advanced Squamous Cell Carcinoma of Head and Neck (HNSCC)
Brief Title: A Study of Dasatinib, Cetuximab and Radiation With or Without Cisplatin in HNSCC
Acronym: Dasatinib
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J08101; CA180123 (Other Grant/Funding Number: BMS)
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Head and Neck Cancer
Keywords: HNSCC; Dasatinib; Cetuximab; Cisplatin
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Dasatinib; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dasatinib/Cetuximab/RT (Experimental): In Cohort A , there will be an initial "run-in period" of single agent cetuximab loading dose of 400mg/m2 on day1, cetuximab maintenance dose 250mg/m2 on day 8 and oral dasatinib at specific dose level from day 8-14.
  Cohort A will consist of patients with AJCC stage II (T2N0) and III (T1-2N1) SCCHN of oral cavity, oropharynx, T2N0 hypopharynx, T2N0-1 supraglottic larynx. Treatment will be dasatinib at specific dose level in combination with cetuximab 250mg/m2 IV and radiation therapy (RT) 70Gy at 2Gy/fn.
  Interventions: Drug: Cetuximab; Drug: Dasatinib; Radiation: Radiation Therapy
- Dasatinib/Cetuximab/cisplatin/RT (Experimental): In Cohort B, there will be an initial "run-in period" of single agent cetuximab loading dose of 400mg/m2 on day1, cetuximab maintenance dose 250mg/m2 on day 8 and oral dasatinib at specific dose level from day 8-14.
  Cohort B will include patients with AJCC stage III (T3N0-1) and IV (T1-4N2-3M0, T4N0-1M0) squamous cell carcinoma of Oral Cavity, Oropharynx, Hypopharynx, and Larynx. Treatment will be daily dasatinib at specific dose level, in combination with q 3 week cisplatin 75mg/m2, weekly cetuximab 250mg/m2 IV and RT 70Gy ( 2gy per fraction).
  Interventions: Drug: Cetuximab; Drug: Dasatinib; Drug: Cisplatin; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Cetuximab — single agent cetuximab loading dose of 400mg/m2 on day1, cetuximab maintenance dose 250mg/m2 on day 8
  Other Names: Erbitux
Drug: Dasatinib — Oral Dasatinib Days 8 through 64.
  Other Names: Sprycel; BMS-354825
Drug: Cisplatin — Q 3 weeks (Days 15, 36 and 57): +/- 3 Days
  Other Names: Cisplatinum; cis-diamminedichloroplatinum(II) (CDDP); Platinol; Platin
  Arms: Dasatinib/Cetuximab/cisplatin/RT
Radiation: Radiation Therapy — Standard Radiation Therapy.

SUMMARY:
Primary Objective for Phase I

1. To determine the maximally tolerated dose (MTD) of daily Oral dasatinib in combination with cetuximab/RT in Cohort A.
2. To determine the MTD of daily oral dasatinib in combination with cisplatin/cetuximab/RT in Cohort B

DETAILED DESCRIPTION:
Primary Objective for Phase I

1. To determine the maximally tolerated dose (MTD) of daily Oral dasatinib in combination with cetuximab/RT in Cohort A, in patients with AJCC stage II (T2N0) and III (T1-2N1) SCCHN of oral cavity, oropharynx, T2N0 hypopharynx, T2N0-1 supraglottic larynx.
2. To determine the MTD of daily oral dasatinib in combination with cisplatin/cetuximab/RT in Cohort B, in patients with AJCC stage III (T3N0-1) and IV (T1-4N2-3M0, T4N0-1M0) squamous cell carcinoma of oral cavity, oropharynx, hypopharynx, and larynx.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically confirmed operable or inoperable squamous cell carcinoma of OC, OP, HP, or larynx prior to proceeding with treatment.
2. Patients must be AJCC stage II (T2N0) or III (T1-2N1) of oral cavity, oropharynx, only T2N0 of hypopharynx, T2N0-1 supraglottic laryngeal cancers (AJCC Fifth Edition, 1997) for Arm A of the study, and must be AJCC stage III (T3N0-1) or IV (T1-4N2-3M0, T4N0-1M0) oral cavity, oropharynx, hypopharynx, glottic and supraglottic laryngeal cancers for Arm B of the study.
3. Patients must have measurable disease,.
4. Subject, age ≥ 18 years.
5. Performance Status (ECOG) 0-1
6. No previous therapy for the tumor, including chemotherapy, radiation therapy, immunotherapy, EGFR targeted therapy, src directed therapies or investigational agents.
7. Adequate Organ Function.

   * Total bilirubin ≤ 1.5 x ULN
   * AST and ALT ≤ 2.5 x ULN
   * Alkaline phosphatase ≤ 2.5 x ULN
   * Hepatic enzymes (AST, ALT) ≤ 2.5 times the institutional ULN.
   * Serum Na, K+, Mg2+, Phosphate and Ca2+ ≥ lower limit of normal (LLN).
   * Serum Creatinine clearance ≥ 60 ml/min.
   * Hemoglobin, neutrophil count, platelets, PT, PTT all Grade 0-1.
   * ANC ≥ 1,500/mL
   * Platelets ≥ 100,000 mL
8. Concomitant medications

   * Patient agrees to discontinue St. Johns Wort, proton pump inhibitors, H2 blockers, aspirin and NSAIDS while receiving dasatinib therapy.
   * Patient agrees that IV and po bisphosphonates will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia.
9. Women of childbearing potential (WOCBP) must have:

   - A negative serum or urine pregnancy test (sensitivity ≤ 25IU HCG/L) within 72 hours prior to the start of study drug administration.
10. Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped.
11. Ability to understand and willingness to sign a written informed consent, including a HIPAA form according to institutional guidelines.

Exclusion Criteria:

1. Any prior radiation above the clavicles
2. Prior head and neck cancer. Any other prior invasive malignancy if disease free interval is ≤ 3 years. Nonmelanomatous carcinomas of the skin and in situ cervical dysplasia are allowed if completely resected within three year interval or can be completely resected prior to starting treatment.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to cetuximab, dasatinib or other agents used in study.
4. Gastrointestinal tract disease resulting in an inability to take or absorb oral or enteral medication.
5. Concurrent medical condition which may increase the risk of toxicity, including:

   * Pleural or pericardial effusion of any grade.
   * Cardiac Symptoms; any of the following should be considered for exclusion:
   * Uncontrolled angina, congestive heart failure or MI within (6 months).
   * Diagnosed congenital long QT syndrome.
   * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes).
   * Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec).
6. Subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to protocol treatment.
7. History of significant bleeding disorder unrelated to cancer, including:

   * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease).
   * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies).
   * Ongoing or recent (≤ 3 months) significant gastrointestinal bleeding.
8. Concomitant Medications, any of the following should be considered for exclusion:

   1. Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib) quinidine, procainamide, disopyramide amiodarone, sotalol, ibutilide, dofetilide erythromycin, clarithromycin chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
   2. The concomitant use of H2 blockers or proton pump inhibitors with dasatinib is not recommended. The use of antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving dasatinib therapy. If antacid therapy is needed, the antacid dose should be administered at least 2 hours prior to or 2 hours after the dose of dasatinib.
9. Patient may not be receiving any prohibited CYP3A4 inhibitors. Refer to section 10 for other concomitant medications you may wish to prohibit based on disease/patient population.
10. Women who:

    * are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug, or
    * have a positive pregnancy test at baseline, or
    * are pregnant or breastfeeding
11. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shanthi Marur, MD, Principal Investigator — Johns Hopkins Universtiy
Locations (2):
- United States (2):
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Ohio State University Medical Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 22 patients were consented. One patient was a screen failure, one patient withdrew consent before initiating any treatment per protocol and patient was replaced in the run-in period before assignment to Cohort A.
Groups:
- Cohort A T2N0, T1-2N1 SCCHN: There will be an initial "run-in period" of single agent cetuximab loading dose of 400mg/m2 on day1, cetuximab maintenance dose 250mg/m2 on day 8 and oral dasatinib from day 8-14.
  Cohort A will consist of patients with AJCC stage II (T2N0) and III (T1-2N1) SCCHN of oral cavity, oropharynx, T2N0 hypopharynx, T2N0-1 supraglottic larynx. Treatment will be dasatinib in combination with cetuximab and radiation therapy (RT).
  Cetuximab: single agent cetuximab loading dose of 400mg/m2 on day1, cetuximab maintenance dose 250mg/m2 on day 8
  Dasatinib: Oral Dasatinib Days 8 through 64.
  Radiation Therapy: Standard Radiation Therapy.
- Cohort B T3N0-1,T1-4N2-3M0, T4N0-1M0 SCCHN: There will be an initial "run-in period" of single agent cetuximab loading dose of 400mg/m2 on day1, cetuximab maintenance dose 250mg/m2 on day 8 and oral dasatinib from day 8-14.
  Cohort B will include patients with AJCC stage III (T3N0-1) and IV (T1-4N2-3M0, T4N0-1M0) squamous cell carcinoma (SCC) of Oral Cavity, Oropharynx, Hypopharynx, and Larynx. Treatment will be daily dasatinib, in combination with q 3 week cisplatin, weekly cetuximab and RT.
  Cetuximab: single agent cetuximab loading dose of 400mg/m2 on day1, cetuximab maintenance dose 250mg/m2 on day 8
  Dasatinib: Oral Dasatinib Days 8 through 64.
  Cisplatin: Q 3 weeks (Days 15, 36 and 57): +/- 3 Days
  Radiation Therapy: Standard Radiation Therapy.
Period: Overall Study
Arm/Group | Cohort A T2N0, T1-2N1 SCCHN | Cohort B T3N0-1,T1-4N2-3M0, T4N0-1M0 SCCHN
Started | 7 | 12
Completed | 6 | 11
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort A: In both Cohort A and B, there will be an initial "run-in period" of single agent cetuximab loading dose of 400mg/m2 on day1, cetuximab maintenance dose 250mg/m2 on day 8 and oral dasatinib from day 8-14.
  Cohort A will consist of patients with AJCC stage II (T2N0) and III (T1-2N1) SCCHN of oral cavity, oropharynx, T2N0 hypopharynx, T2N0-1 supraglottic larynx. Treatment will be dasatinib in combination with cetuximab and radiation therapy (RT).
  Cetuximab: single agent cetuximab loading dose of 400mg/m2 on day1, cetuximab maintenance dose 250mg/m2 on day 8
  Dasatinib: Oral Dasatinib Days 8 through 64.
  Radiation Therapy: Standard Radiation Therapy.
- Cohort B: In both Cohort A and B, there will be an initial "run-in period" of single agent cetuximab loading dose of 400mg/m2 on day1, cetuximab maintenance dose 250mg/m2 on day 8 and oral dasatinib from day 8-14.
  Cohort B will include patients with AJCC stage III (T3N0-1) and IV (T1-4N2-3M0, T4N0-1M0) squamous cell carcinoma of Oral Cavity, Oropharynx, Hypopharynx, and Larynx. Treatment will be daily dasatinib, in combination with q 3 week cisplatin, weekly cetuximab and RT.
  Cetuximab: single agent cetuximab loading dose of 400mg/m2 on day1, cetuximab maintenance dose 250mg/m2 on day 8
  Dasatinib: Oral Dasatinib Days 8 through 64.
  Cisplatin: Q 3 weeks (Days 15, 36 and 57): +/- 3 Days
  Radiation Therapy: Standard Radiation Therapy.
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 7 | 12 | 19
Age, Continuous [Median (Full Range); unit: years] — Age in years collected at screening
  years | 65 [60 to 70] | 58 [48 to 68] | 59 [48 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 9 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 5 | 10 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 12 | 19

OUTCOME MEASURES:

1. Primary Outcome: MTD of Daily Oral Dasatinib in Combination With Cetuximab/RT in Cohort A and Daily Oral Dasatinib in Combination With Cetuximab/Cis or Carboplatin/RT in Cohort B 2. MTD of Daily Oral Dasatinib in Combination With Cisplatin/Cetuximab/RT in Cohort B
Description: The Maximum Tolerated Dose (MTD) for Dasatinib was defined as a) the dose producing DLT ( Dose limiting toxicity) in 0-1 out of 6 patients, or b) the dose level below the dose which produced DLT in <2 out of 6 patients, or c) the dose of 150mg PO QD with less than 33% rate of DLT.
Time Frame: Last day of Radiation
Population: MTD not reached. Data table reports dosage received by each participant. Study closed to slow accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 7 | 12
Participants
  Dose 70 mg | 4 | 7
  Dose 100mg | 3 | 3
  Dose 150mg | 0 | 2

ADVERSE EVENTS:
Time Frame: From start of treatment to 30 days after completion of RT and last dose of Dasatinib. All-cause mortality was based on 2-year follow-up.
Description: This study utilized the Cancer Therapy Evaluation Program Common Toxicity criteria (CTC) version 3.0 for toxicity and event reporting. Dose limiting toxicities were observed until patients completed radiation therapy.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 1/7 | 1/12
Serious Adverse Events (participants affected / at risk) | 1/7 | 5/12
Other Adverse Events (participants affected / at risk) | 7/7 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=7) | Cohort B (N=12)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Grade 2 hypoxia
acute renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) — Grade 3 Pre-renal acute renal failure
dehydration (General disorders) | 0 (0) | 2 (2) — grade 2
Sepsis (General disorders) | 0 (0) | 1 (1) — Grade 2
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Grade 3
hypophosphatemia (General disorders) | 0 (0) | 1 (1) — grade 3
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Grade 2
Febrile neutropenia (Infections and infestations) | 0 (0) | 1 (1) — grade 3
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Grade 3
bacteremia (Infections and infestations) | 0 (0) | 1 (1) — Grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=7) | Cohort B (N=12)
Peg tube site pain (Gastrointestinal disorders) | 6 (6) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (6) | 11 (11)
Vomiting (Gastrointestinal disorders) | 3 (3) | 8 (8)
Constipation (Gastrointestinal disorders) | 5 (5) | 10 (10)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 12 (12)
Fatigue (General disorders) | 5 (5) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 8 (8)
Dysguesia (Gastrointestinal disorders) | 4 (4) | 10 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 5 (7) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 7 (7)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dry mouth (General disorders) | 6 (6) | 8 (8)
Fever (Infections and infestations) | 1 (1) | 5 (5)
oral mucositis (General disorders) | 6 (6) | 11 (11)
elevated AST (Hepatobiliary disorders) | 1 (1) | 1 (1)
elevated ALT (Hepatobiliary disorders) | 1 (1) | 1 (1)
abcess (Infections and infestations) | 1 (1) | 1 (1)
hemetemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
hypophosphatemia (General disorders) | 0 (0) | 2 (2)
hypomagnesemia (General disorders) | 0 (0) | 2 (2)
hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No